CLINICAL TRIAL: NCT06382389
Title: Efficacy of EMONO as an add-on Therapy to Conventional Antidepressants for the Treatment of Depressive Symptoms in Nursing-home Residents With Neurocognitive Disorders: a Randomized Controlled Trial
Brief Title: Efficacy of EMONO as an add-on Therapy to Conventional Antidepressants for the Treatment of Depressive Symptoms in Nursing-home Residents With Neurocognitive Disorders: a Randomized Controlled Trial-
Acronym: PROTO-EHPAD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DR220204; 2023-504691-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Depression; Neurocognitive Disorders
Keywords: Nitrous Oxide
MeSH Terms: conditions — Depression; Neurocognitive Disorders | interventions — Nitrous Oxide; Air

STUDY DESIGN:
Intervention Model Description: Parallel assignement
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMONO (Experimental): Equimolar Mixture of Oxygen and Nitrous Oxide (50%O2 / 50%N2O) Active drug: Nitrous Oxide
  Interventions: Drug: EMONO
- medical air (Active Comparator): Comparator : medical Air (78% N2 / 22% O2)
  Interventions: Drug: Medical air

INTERVENTIONS:
Drug: EMONO — Exposure of Emono via facial mask
  Other Names: Nitrous oxide
  Arms: EMONO
Drug: Medical air — exposure to Medical Air
  Other Names: comparator
  Arms: medical air

SUMMARY:
Depression in neurocognitive disorders (Alzheimers' disease and related disoders) is a highly prevalent condition, especially in nursing homes. While it is associated with significant distress, the current conventional antidepressants have shown only modest efficacy and exposed to potentially severe side effects.

Recent evidence suggests that nitrous oxide (N2O) in its most commonly used packaging of EMONO (Equimolar Mixture of Oxygen and Nitrous Oxide) has rapid antidepressant properties and a good safety profile. However, no study has investigating the antidepressant effect of EMONO in a population of depressed older adults with moderate to severe neurocognitive disorders in nursing homes.

The principal goal of the PROTO-EHPAD study is to compare the changes in depressive symptoms in such individuals in a randomized controlled trial with a follow up period of 8 weeks, with a dosage escalation procedure.

DETAILED DESCRIPTION:
Participants will be exposed to 3 sessions of EMONO (or Medical Air), with intervals of 1 week between sessions : a first session of 20 minutes, a second of 40 minutes one week later and a final session of 60 minutes one week later. Efficacy will be assessed 1 week after each session and 4 weeks after the last session.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 and over living in nursing home
* Diagnosis of major neurocognitive disorder according to DSM-V for at least 6 month
* MMSE <= 20/30
* NPI depression >= 4/12
* Patient, family and legal representive consent where applicable Person affiliated to a social security schem

Exclusion Criteria:

* NPI agitation > 6/12
* Unstable somatic pathology (in particular unstable neurological or cardiological pathologies at risk of interfering with the diffusion of MEOPA) and any unexplained recent neurological abnormality.
* Contraindications to the use of MEOPA
* Patients who have already been treated with MEOPA in the 6 months prior to inclusion, for example for painful treatment
* Sub-physiological plasma vitamin B12 or B9 concentration (below the lower limit of the laboratory value).
* A person participating in a clinical drug study or in a period of exclusion from any clinical study due to previous participation
* Personne participant à une étude clinique médicamenteuse ou en période d'exclusion de toute étude clinique du fait d'une précédente participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes in the CORNELL depression severitý scale between S4 (one week after the last administration of MEOPA or medical air) and S1 (baseline). | baseline, week 4
  The CORNELL is a validated scale specifically designed for depression in major neurocognitive disorders

SECONDARY OUTCOMES:
CORNELL scale and GDS scale at weeks 1, 2, 3, 4 and 8 | baseline, weeks 1, 2, 3, 4 and 8
  The Geriatric Depression Scale is a self assessed scale for depression in older individuals
CGI-S and CGI-I scales at weeks 1, 2, 3, 4 and 8 | baseline, weeks 1, 2, 3, 4 and 8
  CGI assesses the clinical global impression of the clinician
The measurement of well-being by the EVIBE visual analogue scale at weeks 1, 2, 3, 4, and 8 | baseline, weeks 1, 2, 3, 4 and 8
  EVIBE is a visual analog scale specifically designed to measure well being in major cognitive disorders
Collection of adverse events at all study visits | baseline, weeks 1, 2, 3, 4 and 8
  any adverse events will be collected

IPD SHARING:
Plan to Share IPD: No